CLINICAL TRIAL: NCT06854601
Title: A Multicenter, Double-blind, Randomized, Placebo-controlled Clinical Trial in Three Parallel Groups to Evaluate the Effectiveness and Safety of Mexidol® Film-coated Tablets, 125 mg (LLC 'NPK PHARMASOFT', Russia) in the Treatment of Attention Deficit Hyperactivity Disorder (ADHD) in Children Aged 6-12 Years With Various Dosing Regimens (MEGA).
Brief Title: Safety and Efficacy of Mexidol® for ADHD in Children Aged 6-12
Acronym: MEGA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pharmasoft (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MexidolMEGA2020; PHS-ADHD-002-MEX-TAB (Other: Pharmasoft)
Record Dates: First submitted 2025-02-11; First posted 2025-03-03 (Actual); Results first posted 2025-08-17 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-07

CONDITIONS: Attention Deficit Hyperactivity Disorder (ADHD); Anxiety Disorders and Symptoms
Keywords: Mexidol; hyperactivity; ADHD; oppositional defiant disorder; inattention; Neurodevelopmental disorders; Hyperactive behavior; Impulsive behavior; anxiety
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Anxiety Disorders; Spasm; Oppositional Defiant Disorder; Neurodevelopmental Disorders; Impulsive Behavior | interventions — emoxypine succinate

STUDY DESIGN:
Intervention Model Description: Multicenter, double-blind, randomized, placebo-controlled clinical trial in three parallel groups to evaluate efficacy and safety
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Main (Mexidol) + Control (Placebo) (Other): Participants received Mexidol 125 mg 1 tablet orally once a day and Mexidol Placebo matching Mexidol 125 mg 1 tablet orally once a day for 42 days.
  Interventions: Drug: Mexidol + Placebo
- Main (Mexidol) (Active Comparator): Participants received Mexidol 125 mg 1 tablet orally twice a day for 42 days.
  Interventions: Drug: Mexidol
- Control (Placebo) (Placebo Comparator): Participants received Mexidol Placebo matching Mexidol 125 mg 1 tablet orally twice a day for 42 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Mexidol — 125 mg tablets
  Arms: Main (Mexidol)
Drug: Placebo — Placebo tablets
  Arms: Control (Placebo)
Drug: Mexidol + Placebo — Combination of Mexidol and Placebo
  Arms: Main (Mexidol) + Control (Placebo)

SUMMARY:
The primary objective of this study was to evaluate the efficacy and safety of Mexidol® film-coated tablets (125 mg) compared to a placebo in children aged 6 to 12 years with Attention Deficit Hyperactivity Disorder (ADHD). This multicenter, prospective, double-blind, randomized trial included 333 children who met the diagnostic criteria established by the International Classification of Diseases (ICD-10) and the Diagnostic and Statistical Manual of Mental Disorders (DSM-5). Participants received either Mexidol or placebo for 42 days, and various efficacy and safety parameters were assessed.

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent for participation in the study from the patient's parents.
2. Patients - boys and girls aged 6 to 12 years, inclusive, at the time of signing the informed consent.
3. The child is raised by a father and/or mother.
4. The child is attending general education preschool or school institutions.
5. Diagnosis of Attention Deficit Hyperactivity Disorder (ADHD) established in accordance with ICD-10 and DSM-5 criteria by a psychiatrist or neurologist, specifically:

   - According to DSM-5:
   1. Six or more symptoms of inattention persisting for at least 6 months and/or
   2. Six or more symptoms of hyperactivity and impulsivity persisting for at least 6 months
   3. Symptoms are present in at least two areas of functioning (in preschool or school and at home).

      - And/or according to ICD-10:
   4. Presence of at least 6 symptoms of inattention
   5. Presence of at least 3 symptoms of hyperactivity
   6. Presence of at least 1 symptom of impulsivity
   7. Persisting for at least 6 months.
6. Moderate severity of ADHD as determined by the Clinical Global Impression - Severity Scale for ADHD (CGI-ADHD-S), not requiring hospitalization for treatment.
7. No more than two comorbid disorders that do not require additional pharmacotherapy, in the investigator's opinion, during the study period.

Exclusion Criteria:

Individuals who exhibit at least one of the following characteristics were not included in the study:

1. Increased sensitivity to the active substance of the investigational drug (ethylmethylhydroxypyridine succinate) and/or other components of the drug.
2. Liver dysfunction: ALT and/or AST ≥2.5 times the upper limit of normal (ULN) based on screening lab results.
3. Kidney dysfunction: serum creatinine ≥1.5 times ULN based on screening lab results.
4. Intracranial pathology (including but not limited to: intracranial hemorrhage, tumors, infections, history of head trauma, excluding concussion).
5. Co-occurring autism spectrum disorders, Asperger syndrome.
6. Intellectual disability of any degree.
7. Other mental disorders, except for behavioral disorders (ICD-10 code F91).
8. Inability to discontinue psychotropic medications used for the treatment of ADHD.
9. Other somatic and/or neurological disorders requiring treatment with medications that may affect the efficacy of the investigational drug (including but not limited to: epilepsy, depression).
10. Use of nootropic, vasoactive medications, neuroprotectors, antioxidants, or metabolic agents within 7 days or 5 half-lives (whichever is longer) prior to randomization.
11. Presence of any oncological disease in the medical history within 5 years prior to the screening visit.
12. Participation in any other clinical study of drugs and/or medical devices within 3 months prior to the screening visit and/or 5 half-lives, whichever is longer.
13. Inability or unwillingness to comply with protocol requirements, including for physical, mental, or social reasons, in the opinion of the investigator.
14. Lactose intolerance, lactase deficiency, glucose-galactose malabsorption.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 333 (Actual)
Dates: Start 2019-07-13 (Actual); Primary Completion 2020-07-13 (Actual); Study Completion 2020-07-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Polina S. Nikiforova, MD, Principal Investigator — State Autonomous Healthcare Institution of the Sverdlovsk Region "Multispecialty Clinical Medical Center 'Bonum'; Nikolay N. Zavadenko, Dr.Med.Sci, Prof., Principal Investigator — Federal State Autonomous Educational Institution of Higher Education "Russian National Research Medical University named after N.I. Pirogov" Ministry of Health of the Russian Federation; Olga V. Khaletskaya, Dr.Med.Sci, Prof., Principal Investigator — Limited Liability Company "NizhMedClinic"; Elena V. Levitina, Dr.Med.Sci, Prof., Principal Investigator — Federal State Budgetary Educational Institution of Higher Education "Tyumen State Medical University" Ministry of Health of the Russian Federation,; Irina N. Vakula, MD, Principal Investigator — Limited Liability Company "Center for Professional Therapy"; Olga S. Panina, Cand.Med.Sci, MD, Principal Investigator — Limited Liability Company "DNA Research Center"; Dina D. Gainetdinova, Dr.Med.Sci, Prof., Principal Investigator — Federal State Budgetary Educational Institution of Higher Education "Kazan State Medical University" Ministry of Health of the Russian Federation; Anna N. Platonova, Cand.Med.Sci, MD, Principal Investigator — State Budgetary Healthcare Institution of the City of Moscow "Scientific and Practical Center for Child Psychoneurology of the Moscow Department of Healthcare"; Yuliya O. Boychevskaya, MD, Principal Investigator — State Budgetary Healthcare Institution "Specialized Clinical Psychiatric Hospital №1" of the Ministry of Health of the Krasnodar Territory; Natalya E. Maksimova, Cand.Med.Sci, MD, Principal Investigator — Federal State Budgetary Educational Institution of Higher Education "Tver State Medical University" Ministry of Health of the Russian Federation; Elena M. Kryukova, MD, Principal Investigator — State Budgetary Healthcare Institution "Orenburg Regional Clinical Psychiatric Hospital №1"; Elmira S. Sagutdinova, Cand.Med.Sci, MD, Principal Investigator — Limited Liability Company "European Medical Center 'UGMK-Health'"; Anna S. Nezabudkina, MD, Principal Investigator — Limited Liability Company "Medical Technologies"; Viktor V. Mashin, Dr.Med.Sci, Prof., Principal Investigator — State Healthcare Institution "Central Clinical Medical-Sanitary Unit named after Honored Doctor of Russia V.A. Egorov"
Locations (14):
- Russia (14):
  - State Autonomous Healthcare Institution of the Sverdlovsk Region "Multispecialty Clinical Medical Center 'Bonum', Yekaterinburg, Ural Region
  - Federal State Budgetary Educational Institution of Higher Education "Kazan State Medical University" Ministry of Health of the Russian Federation, Kazan'
  - State Budgetary Healthcare Institution "Specialized Clinical Psychiatric Hospital №1" of the Ministry of Health of the Krasnodar Territory, Krasnodar
  - Limited Liability Company "Center for Professional Therapy", Krasnodar
  - Federal State Autonomous Educational Institution of Higher Education "Russian National Research Medical University named after N.I. Pirogov" Ministry of Health of the Russian Federation, Moscow
  - State Budgetary Healthcare Institution of the City of Moscow "Scientific and Practical Center for Child Psychoneurology of the Moscow Department of Healthcare", Moscow
  - Limited Liability Company "NizhMedClinic", Nizhny Novgorod
  - State Budgetary Healthcare Institution "Orenburg Regional Clinical Psychiatric Hospital №1", Orenburg
  - Limited Liability Company "Medical Technologies", Saint Petersburg
  - Limited Liability Company "DNA Research Center", Saratov
  - Federal State Budgetary Educational Institution of Higher Education "Tver State Medical University" Ministry of Health of the Russian Federation, Tver'
  - Federal State Budgetary Educational Institution of Higher Education "Tyumen State Medical University" Ministry of Health of the Russian Federation, Tyumen
  - State Healthcare Institution "Central Clinical Medical-Sanitary Unit named after Honored Doctor of Russia V.A. Egorov", Ulyanovsk
  - Limited Liability Company "European Medical Center 'UGMK-Health'", Yekaterinburg

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited based on protocol requirements at 14 clinical sites between July 2019 and May 2020. The first participant was enrolled on 13 July, 2019 and the last participant was enrolled on 22 May, 2020.
Pre-assignment Details: Of 340 screened participants, 333 met inclusion criteria and were randomized to treatment.
Period: Overall Study
Arm/Group | Main (Mexidol) + Control (Placebo) | Main (Mexidol) | Control (Placebo)
Started | 111 | 111 | 111
Completed | 111 | 111 | 110
Not Completed | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Main (Mexidol) + Control (Placebo) | Main (Mexidol) | Control (Placebo) | Total
Number analyzed (Participants) | 111 | 111 | 111 | 333
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 111 | 111 | 111 | 333
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Median (Inter-Quartile Range); unit: Years] | 8 [7 to 10] | 9 [7 to 10] | 8 [7 to 10] | 8 [7 to 10]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 29 | 31 | 97
  Male | 74 | 82 | 80 | 236
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: Participants]
  Russia | 111 | 111 | 111 | 333
SNAP-IV, Subscales "Inattention" and "Hyperactivity/Impulsivity" at Visit 2 (Randomization Visit) [Mean (Standard Deviation); unit: score on a scale] — The Swanson, Nolan and Pelham Teacher and Parent Rating Scale (SNAP-IV) is a 90-question self-report inventory designed to measure attention deficit hyperactivity disorder and oppositional defiant disorder symptoms in children and young adults. The SNAP-IV is based on a 0 to 3 rating scale: Not at all = 0, Just a little = 1, Often = 2, and Very often = 3. The questions measure different domains of ADHD and ODD. Subscale scores are calculated by summing the scores on the subset and dividing by the number of items in the subset. Higher score indicates higher symptom severity.
  score on a scale | 32.72 (6.73) | 32.37 (6.91) | 33.03 (7.18) | 32.70 (6.93)
SNAP-IV, Subscale "Inattention" at Visit 1 (Screening) [Mean (Standard Deviation); unit: score on a scale] — The Swanson, Nolan and Pelham Teacher and Parent Rating Scale (SNAP-IV) is a 90-question self-report inventory designed to measure different domains of ADHD and ODD. The SNAP-IV is based on a 0 to 3 rating scale: Not at all = 0, Just a little = 1, Often = 2, and Very often = 3. Subscale scores on the SNAP-IV are calculated by summing the scores on the subset and dividing by the number of items in the subset. Higher score indicates higher symptom severity.
  score on a scale | 17.84 (3.52) | 17.38 (3.79) | 18.00 (3.76) | 17.74 (3.69)
SNAP-IV, Subscale "Hyperactivity/Impulsivity at Visit 1 (Screening) [Mean (Standard Deviation); unit: score on a scale] — The Swanson, Nolan and Pelham Teacher and Parent Rating Scale (SNAP-IV) is a 90-question self-report inventory designed to measure different domains of ADHD and ODD. The SNAP-IV is based on a 0 to 3 rating scale: Not at all = 0, Just a little = 1, Often = 2, and Very often = 3. Subscale scores on the SNAP-IV are calculated by summing the scores on the subset and dividing by the number of items in the subset. Higher score indicates higher symptom severity.
  score on a scale | 14.88 (4.27) | 14.99 (4.22) | 15.03 (4.51) | 14.96 (4.32)
SNAP-IV, Subscale "Oppositional Defiant Disorder" at Visit 1 (Screening) [Mean (Standard Deviation); unit: score on a scale] — The Swanson, Nolan and Pelham Teacher and Parent Rating Scale (SNAP-IV) is a 90-question self-report inventory designed to measure different domains of ADHD and ODD. The SNAP-IV is based on a 0 to 3 rating scale: Not at all = 0, Just a little = 1, Often = 2, and Very often = 3. Subscale scores on the SNAP-IV are calculated by summing the scores on the subset and dividing by the number of items in the subset. Higher score indicates higher symptom severity.
  score on a scale | 5.16 (5.42) | 4.64 (5.62) | 5.24 (4.97) | 5 (5.33)
SNAP-IV, Subscale "Connors Index" at Visit 1 (Screening) [Mean (Standard Deviation); unit: score on a scale] — The Swanson, Nolan and Pelham Teacher and Parent Rating Scale (SNAP-IV) is a 90-question self-report inventory designed to measure different domains of ADHD and ODD. The SNAP-IV is based on a 0 to 3 rating scale: Not at all = 0, Just a little = 1, Often = 2, and Very often = 3. Subscale scores on the SNAP-IV are calculated by summing the scores on the subset and dividing by the number of items in the subset. Higher score indicates higher symptom severity.
  score on a scale | 12.03 (5.11) | 11.39 (5.36) | 12.33 (5.43) | 11.92 (5.30)
SCAS-Parent at Visit 2 (Randomization Visit) [Mean (Standard Deviation); unit: score on a scale] — The Spence Children's Anxiety Scale - Parent Version (SCAS-Parent) is a 39-item parent report measure designed to assess anxiety symptoms in children. It evaluates six distinct domains of anxiety that align with clinical diagnostic categories. Each question addresses the frequency of certain anxiety symptoms, measured on a 0-3 scale from "never", "sometimes", "often", to "always". SCAS-Parent scores consist of a total raw score (range from 0 to 114) and six sub-scale scores, with higher scores indicating greater severity of anxiety symptoms.
  score on a scale | 13.13 (14.84) | 13.27 (15.36) | 13.27 (13.63) | 13.22 (14.58)
ADHD-RS-IV at Visit 2 (Randomization Visit) [Mean (Standard Deviation); unit: score on a scale] — The Attention Deficit Hyperactivity Disorder Rating Scale (ADHD-RS) is an 18-question inventory used to aid in the diagnosis of attention deficit hyperactivity disorder (ADHD) in children. Each question measures the frequency of the behavior on a 0-3 scale from "rarely or never", "sometimes", "often", to "very often". The questionnaire is intended to be filled out by parents and teachers. Higher scores indicate greater severity of ADHD symptoms.
  score on a scale | 32.55 (6.92) | 32.68 (6.90) | 32.77 (6.88) | 32.66 (6.88)
CGI-ADHD-S Scale before treatment [Count of Participants; unit: Participants] — The Clinical Global Impressions-ADHD-Severity (CGI-ADHD-S) is a clinician-rated scale used to assess the severity of Attention Deficit Hyperactivity Disorder (ADHD) symptoms. This tool is part of the Clinical Global Impressions (CGI) scales. It typically consists of a single item that rates the severity of ADHD on a 7-point scale: 1=normal, not at all ill; 2=borderline mentally ill; 3=mildly ill; 4=moderately ill; 5=markedly ill; 6=severely ill; 7=among the most extremely ill patients.
  Participants
    Level 2 (borderline mentally ill) | 0 | 0 | 0 | 0
    Level 3 (mildly ill) | 0 | 0 | 0 | 0
    Level 4 (moderately ill) | 111 | 111 | 111 | 333
    Level 5 (markedly ill) | 0 | 0 | 0 | 0
PedMIDAS at Visit 2 (Randomization Visit) [Mean (Standard Deviation); unit: days] — The Pediatric Migraine DisabilityAssessment (PedMIDAS) questionnaire is used toassess the impact of headaches on schoolperformance (three questions), activities at home (onequestion on homework or chores), and social and/orsports functions (two questions). It is scored bysumming the answers across the six questions.PedMIDAS score range from 0 to 10 indicates little tonone disability grade, score range from 11 to 30indicates mild disability grade, score range from 31 to50 indicates moderate disability grade and score rangegreater than 50 indicates severe disability grade. Population: The scoreson this questionnaire were evaluated only for patientswho were found to have a headache. Thus, the data forcomparing the results at the end of the therapy with theresults at the beginning of the therapy were availablefor 18 patients.
  days
    Number of days with limited daily activities: number analyzed (Participants) | 8 | 3 | 7 | 18
    Number of days with limited daily activities | 10.96 (19.76) | 0.56 (0.51) | 1.62 (1.82) | 5.59 (13.66)
    Number of days with a headache: number analyzed (Participants) | 8 | 3 | 7 | 18
    Number of days with a headache | 9.04 (10.52) | 3.22 (2.27) | 4.86 (2.30) | 6.44 (7.35)
PedMIDAS at Visit 2 (Randomization Visit) [Mean (Standard Deviation); unit: scores on ascale] — The Pediatric Migraine DisabilityAssessment (PedMIDAS) questionnaire is used toassess the impact of headaches on schoolperformance (three questions), activities at home (onequestion on homework or chores), and social and/orsports functions (two questions). It is scored bysumming the answers across the six questions.PedMIDAS score range from 0 to 10 indicates little tonone disability grade, score range from 11 to 30indicates mild disability grade, score range from 31 to50 indicates moderate disability grade and score rangegreater than 50 indicates severe disability grade. Population: The scoreson this questionnaire were evaluated only for patientswho were found to have a headache. Thus, the data forcomparing the results at the end of the therapy with theresults at the beginning of the therapy were availablefor 18 patients.
  scores on ascale
    Moderate headache severity: number analyzed (Participants) | 8 | 3 | 7 | 18
    Moderate headache severity | 4.25 (2.19) | 3.00 (1.00) | 3.86 (1.68) | 3.89 (1.81)
    Maximal headache severity: number analyzed (Participants) | 8 | 3 | 7 | 18
    Maximal headache severity | 5.75 (2.19) | 4.00 (0.00) | 6.14 (2.12) | 5.61 (2.03)

OUTCOME MEASURES:

1. Primary Outcome: The Average Change in the Total Score Across the "Inattention" and "Hyperactivity/Impulsivity" Subscales of the Swanson, Nolan and Pelham Teacher and Parent Rating Scale (SNAP-IV) After 6 Weeks of Therapy Compared to the Baseline Level.
Description: The Swanson, Nolan and Pelham Teacher and Parent Rating Scale (SNAP-IV) is a 90-question self-report inventory designed to measure attention deficit hyperactivity disorder and oppositional defiant disorder symptoms in children and young adults. The SNAP-IV is based on a 0 to 3 rating scale: Not at all = 0, Just a little = 1, Often = 2, and Very often = 3. The questions measure different domains of ADHD and ODD. Subscale scores are calculated by summing the scores on the subset and dividing by the number of items in the subset. The main criterion for the treatment efficacy was the mean change in the total score on the "inattention" and "hyperactivity/impulsivity" subscales after 6 weeks of therapy. A conclusion of superiority of Mexidol over placebo can be made if the upper limit of the 95% confidence interval for the difference in mean changes is negative. 55 point scale: min value 0, max value 54, higher scores mean a worse outcome.
Time Frame: Visit 5 (after 6 weeks of therapy) compared to the baseline level (Visit 2 Day 1 = Randomization Visit)
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Main (Mexidol) + Control (Placebo) | Main (Mexidol) | Control (Placebo)
Number analyzed (Participants) | 111 | 111 | 111
score on a scale
  SNAP-IV at Visit 5 | 25.41 [23.91 to 26.92] | 23.04 [21.49 to 24.58] | 29.10 [27.66 to 30.54]
  Difference at Visit 5 compared to Visit 2 | -7.31 [-8.44 to -6.17] | -9.33 [-10.59 to -8.07] | -3.93 [-5.11 to -2.75]

2. Secondary Outcome: Average Change in the the Swanson, Nolan and Pelham Teacher and Parent Rating Scale (SNAP-IV), Subscale "Inattention"
Description: The Swanson, Nolan and Pelham Teacher and Parent Rating Scale (SNAP-IV) is a 90-question self-report inventory designed to measure attention deficit hyperactivity disorder (ADHD) and oppositional defiant disorder (ODD) symptoms in children and young adults. The SNAP-IV is based on a 0 to 3 rating scale: Not at all = 0, Just a little = 1, Often = 2, and Very often = 3. The questions measure different domains of ADHD and ODD. Subscale scores on the SNAP-IV are calculated by summing the scores on the subset and dividing by the number of items in the subset. The score for any subset is expressed as the Average Rating-Per-Item. 28 point scale: min value 0, max value 27, higher scores mean a worse outcome.
Time Frame: Visit 5 (after 6 weeks of therapy) compared to the baseline level (Visit 1 Day 0 = Screening)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Main (Mexidol) + Control (Placebo) | Main (Mexidol) | Control (Placebo)
Number analyzed (Participants) | 111 | 111 | 111
score on a scale
  SNAP-IV, Subscale "Inattention" at Visit 5 | 14.04 (3.79) | 12.84 (4.50) | 15.95 (3.85)
  Difference at Visit 5 compared to Visit 1 | -3.80 (3.62) | -4.54 (3.87) | -2.05 (3.55)

3. Secondary Outcome: Average Change in the Swanson, Nolan and Pelham Teacher and Parent Rating Scale (SNAP-IV), Subscale "Hyperactivity/Impulsivity"
Description: as for outcome 2
Time Frame: Visit 5 (after 6 weeks of therapy) compared to the baseline level (Visit 1 Day 0 = Screening)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Main (Mexidol) + Control (Placebo) | Main (Mexidol) | Control (Placebo)
Number analyzed (Participants) | 111 | 111 | 111
score on a scale
  SNAP-IV, Subscale "Hyperactivity/Impulsivity" at Visit 5 | 11.38 (5.06) | 10.20 (4.58) | 13.15 (4.76)
  Difference at Visit 5 compared to Visit 1 | -3.50 (3.36) | -4.79 (3.64) | -1.87 (3.28)

4. Secondary Outcome: Average Change in the Swanson, Nolan and Pelham Teacher and Parent Rating Scale (SNAP-IV), Subscale "Oppositional Defiant Disorder"
Description: The Swanson, Nolan and Pelham Teacher and Parent Rating Scale (SNAP-IV) is a 90-question self-report inventory designed to measure attention deficit hyperactivity disorder (ADHD) and oppositional defiant disorder (ODD) symptoms in children and young adults. The SNAP-IV is based on a 0 to 3 rating scale: Not at all = 0, Just a little = 1, Often = 2, and Very often = 3. The questions measure different domains of ADHD and ODD. Subscale scores on the SNAP-IV are calculated by summing the scores on the subset and dividing by the number of items in the subset. The score for any subset is expressed as the Average Rating-Per-Item. 25 point scale: min value 0, max value 24, higher scores mean a worse outcome.
Time Frame: Visit 5 (after 6 weeks of therapy) compared to the baseline level (Visit 1 Day 0 = Screening)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Main (Mexidol) + Control (Placebo) | Main (Mexidol) | Control (Placebo)
Number analyzed (Participants) | 111 | 111 | 111
score on a scale
  SNAP-IV, Subscale "Oppositional Defiant Disorder" at Visit 5 | 4.06 (4.91) | 3.69 (4.88) | 4.43 (4.48)
  Difference at Visit 5 compared to Visit 1 | -1.10 (2.50) | -0.95 (2.57) | -0.81 (2.78)

5. Secondary Outcome: Average Change in the Swanson, Nolan and Pelham Teacher and Parent Rating Scale (SNAP-IV), Subscale "Connors Index"
Description: The Swanson, Nolan and Pelham Teacher and Parent Rating Scale (SNAP-IV) is a 90-question self-report inventory designed to measure attention deficit hyperactivity disorder (ADHD) and oppositional defiant disorder (ODD) symptoms in children and young adults. The SNAP-IV is based on a 0 to 3 rating scale: Not at all = 0, Just a little = 1, Often = 2, and Very often = 3. The questions measure different domains of ADHD and ODD. Subscale scores on the SNAP-IV are calculated by summing the scores on the subset and dividing by the number of items in the subset. The score for any subset is expressed as the Average Rating-Per-Item. 31 point scale: min value 0, max value 30, higher scores mean a worse outcome.
Time Frame: Visit 5 (after 6 weeks of therapy) compared to the baseline level (Visit 1 Day 0 = Screening)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Main (Mexidol) + Control (Placebo) | Main (Mexidol) | Control (Placebo)
Number analyzed (Participants) | 111 | 111 | 111
score on a scale
  SNAP-IV), Subscale "Connors Index" at Visit 5 | 8.71 (4.83) | 8.21 (5.39) | 10.33 (4.57)
  Difference at Visit 5 compared to Visit 1 | -3.32 (2.99) | -3.18 (3.17) | -2.00 (3.37)

6. Secondary Outcome: Average Change in the Spence Children's Anxiety Scale - Parent Version (SCAS-Parent) Score
Description: The Spence Children's Anxiety Scale - Parent Version (SCAS-Parent) is a 39-item parent report measure designed to assess anxiety symptoms in children. Built upon contemporary diagnostic frameworks, the SCAS-Parent evaluates six distinct domains of anxiety that align with clinical diagnostic categories. Each question on the test addresses the frequency of certain anxiety symptoms, measured on a 0-3 scale from "never", "sometimes", "often", to "always". SCAS-Parent scores consist of a total raw score (range from 0 to 114) and six sub-scale scores, with higher scores indicating greater severity of anxiety symptoms. 124 point scale: min value 0, max value 123, higher scores mean a worse outcome.
Time Frame: Visit 5 (after 6 weeks of therapy) compared to the baseline level (Visit 2 Day 1 = Randomization Visit)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Main (Mexidol) + Control (Placebo) | Main (Mexidol) | Control (Placebo)
Number analyzed (Participants) | 111 | 111 | 111
score on a scale
  SCAS-Parent at Visit 5 | 10.23 (13.66) | 10.41 (15.33) | 10.22 (10.64)
  Difference at Visit 5 compared to Visit 2 | -2.90 (5.45) | -2.86 (6.27) | -3.05 (6.76)

7. Secondary Outcome: Average Change in the Attention Deficit Hyperactivity Disorder Rating Scale-IV (ADHD-RS-IV) Score
Description: The Attention Deficit Hyperactivity Disorder Rating Scale (ADHD-RS) is an 18-question inventory used to aid in the diagnosis of attention deficit hyperactivity disorder (ADHD) in children. Each question measures the frequency of the behavior on a 0-3 scale from "rarely or never", "sometimes", "often", to "very often". The questionnaire is intended to be filled out by parents and teachers. Higher scores indicate greater severity of ADHD symptoms. 55 point scale: min value 0, max value 54, higher scores mean a worse outcome.
Time Frame: Visit 5 (after 6 weeks of therapy) compared to the baseline level (Visit 2 Day 1 = Randomization Visit)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Main (Mexidol) + Control (Placebo) | Main (Mexidol) | Control (Placebo)
Number analyzed (Participants) | 111 | 111 | 111
score on a scale
  ADHD-RS-IV at Visit 5 | 25.23 (8.01) | 23.14 (8.26) | 28.85 (7.68)
  Difference at Visit 5 compared to Visit 2 | -7.32 (6.15) | -9.54 (6.88) | -3.92 (6.16)

8. Secondary Outcome: Assessment Using the Clinical Global Impressions for Attention Deficit Hyperactivity Disorder Severity (CGI-ADHD-S) Scale
Description: The Clinical Global Impressions-ADHD-Severity (CGI-ADHD-S) is a clinician-rated scale used to assess the severity of Attention Deficit Hyperactivity Disorder (ADHD) symptoms. This tool is part of the Clinical Global Impressions (CGI) scales. It typically consists of a single item that rates the severity of ADHD on a 7-point scale, ranging from 1 (normal, not at all ill) to 7 (among the most extremely ill patients). 7 point scale: min value 1, max value 7, higher scores mean a worse outcome.
Time Frame: Visit 5 (after 6 weeks of therapy) compared to the baseline level (Visit 2 Day 1 = Randomization Visit)
Measure: Count of Participants; unit: Participants
Arm/Group | Main (Mexidol) + Control (Placebo) | Main (Mexidol) | Control (Placebo)
Number analyzed (Participants) | 111 | 111 | 111
Participants
  Level 2 (borderline mentally ill) | 8 | 8 | 2
  Level 3 (mildly ill) | 26 | 58 | 23
  Level 4 (moderately ill) | 77 | 44 | 86
  Level 5 (markedly ill) | 0 | 1 | 0

9. Secondary Outcome: Assessment Using the Clinical Global Impressions Scale for Improvement (CGI-I)
Description: The Clinical Global Impressions (CGI) Scale is a standardized assessment tool used to rate the severity of illness, change over time, and efficacy of medication. It consists of 3 subscales. The subscale Clinical Global Impression-Improvement (CGI-I) is a 7-point scale that assesses how much the patient's illness has improved or worsened relative to a baseline state at the beginning of the intervention, and rated as: 1, very much improved; 2, much improved; 3, minimally improved; 4, no change; 5, minimally worse; 6, much worse; or 7, very much worse. 7 point scale: min value 1, max value 7, higher scores mean a worse outcome.
Time Frame: Visit 5 (after 6 weeks of therapy) compared to the baseline level (before treatment)
Measure: Count of Participants; unit: Participants
Arm/Group | Main (Mexidol) + Control (Placebo) | Main (Mexidol) | Control (Placebo)
Number analyzed (Participants) | 111 | 111 | 111
Participants
  1, very much improved | 3 | 13 | 2
  2, much improved | 20 | 45 | 10
  3, minimally improved | 61 | 37 | 38
  4, no change | 27 | 14 | 58
  5, minimally worse | 0 | 1 | 3
  6, much worse | 0 | 1 | 0
  7, very much worse | 0 | 0 | 0

10. Secondary Outcome: Assessment Using the Pediatric Migraine Disability Assessment Questionnaire (PedMIDAS), Days
Description: The Pediatric Migraine Disability Assessment questionnaire (PedMIDAS) is used to assess the impact of headaches on school performance (three questions), activities at home (one question on homework or chores), and social and/or sports functions (two questions). The PedMIDAS is scored by summing the answers across the six questions. The frequency and severity are not scored but can be used for clinical reference. PedMIDAS score range from 0 to 10 indicates little to none disability grade, score range from 11 to 30 indicates mild disability grade, score range from 31 to 50 indicates moderate disability grade and score range greater than 50 indicates severe disability grade. Min value 0, max value 240, higher scores mean a worse outcome.
Time Frame: Visit 5 (after 6 weeks of therapy) compared to the baseline level (Visit 2 Day1 = Randomization Visit)
Population: The scores on this questionnaire were evaluated only for patients who were found tohave a headache. Thus, the data for comparing the results at the end of the therapy withthe results at the beginning of the therapy were available for 18 patients.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Main (Mexidol) + Control (Placebo) | Main (Mexidol) | Control (Placebo)
Number analyzed (Participants) | 8 | 3 | 7
days
  Number of days with limited daily activities | 4.25 (10.97) | 0.22 (0.38) | 2.38 (2.03)
  No of days with limited activity: Visit 5 compared to Visit 2 | -6.71 (11.77) | -0.33 (0.33) | 0.76 (1.46)
  Number of days with a headache | 9.58 (10.73) | 5.11 (2.52) | 4.95 (2.52)
  No of days with headache: Visit 5 compared to Visit 2 | 0.54 (8.45) | 1.89 (4.72) | 0.10 (3.72)

11. Secondary Outcome: Assessment Using the Pediatric Migraine Disability Assessment Questionnaire (PedMIDAS), Headache Severity
Description: as for outcome 10
Time Frame: Visit 5 (after 6 weeks of therapy) compared to the baseline level (Visit 2 Day1 = Randomization Visit)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Main (Mexidol) + Control (Placebo) | Main (Mexidol) | Control (Placebo)
Number analyzed (Participants) | 8 | 3 | 7
score on a scale
  Moderate headache severity | 3.88 (2.10) | 3.00 (1.00) | 3.71 (1.25)
  Moderate headache: Visit 5 compared to Visit 2 | -0.38 (1.19) | 0.00 (0.00) | -0.14 (0.90)
  Maximal headache severity | 6.13 (3.00) | 5.33 (2.31) | 5.57 (1.51)
  Max headache: Visit 5 compared to Visit 2 | 0.38 (1.85) | 1.33 (2.31) | -0.57 (1.72)

ADVERSE EVENTS:
Time Frame: From Day 1 (Visit 2) to Day 50+3 (Visit 6) or Early Termination Visit
Arm/Group | Main (Mexidol) + Control (Placebo) | Main (Mexidol) | Control (Placebo)
All-Cause Mortality (participants affected / at risk) | 0/111 | 0/111 | 0/111
Serious Adverse Events (participants affected / at risk) | 0/111 | 1/111 | 1/111
Other Adverse Events (participants affected / at risk) | 14/111 | 26/111 | 20/111
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Main (Mexidol) + Control (Placebo) (N=111) | Main (Mexidol) (N=111) | Control (Placebo) (N=111)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Furuncle (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Main (Mexidol) + Control (Placebo) (N=111) | Main (Mexidol) (N=111) | Control (Placebo) (N=111)
Abdominal pain upper (Gastrointestinal disorders) | 1 (2) | 2 (2) | 0 (0)
Irritable bowel syndrome (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2) | 2 (2) | 2 (2)
Respiratory tract infection (Infections and infestations) | 2 (2) | 2 (2) | 4 (4)
Nasopharyngitis (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Otosalpingitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Rhinitis (Infections and infestations) | 1 (1) | 4 (4) | 3 (3)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Furuncle (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)
Oral allergy syndrome (Immune system disorders) | 0 (0) | 0 (0) | 1 (1)
Seasonal allergy (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 3 (4) | 2 (2)
Disturbance in attention (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Meibomianitis (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Urine abnormality (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Leukocyturia (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Affect lability (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Listless (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Inappropriate affect (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Animal bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2019-10-15): https://cdn.clinicaltrials.gov/large-docs/01/NCT06854601/Prot_000.pdf
  • Statistical Analysis Plan (2019-09-27): https://cdn.clinicaltrials.gov/large-docs/01/NCT06854601/SAP_001.pdf